CLINICAL TRIAL: NCT05547932
Title: The Effect of Ultrasound-guided Rhomboid Intercostal Block and Serratus Anterior Plane Block on Postoperative Respiratory Functions and Analgesia After Breast Surgery
Brief Title: The Effect of Rhomboid Intercostal Block and Serratus Anterior Plane Block on Postoperative Respiratory Functions
Acronym: RIBSAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Başak Altıparmak, Associated Prof Dr, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MSK8/22
Record Dates: First submitted 2022-08-10; First posted 2022-09-21 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Postoperative Pain; Respiratory Function Impaired
Keywords: Analgesia; postoperative pain; rhomboid intercostal block; serratus anterior plane block; respiratory function
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Respiratory Insufficiency; Agnosia; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients will be under general anesthesia and will not know if they received a block procedure or not.
  The investigator, the data collector and the outcome assessor will be completely blind to the study groups. Only the care provider who will perform the block procedures will know the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block Group (Experimental): After endotracheal intubation, patients will be positioned in lateral decubitus position. A linear ultrasound probe will be placed at the edge of scapula at the level of T5-T6. Under sterile conditions, the landmark points (rhomboid major muscle, 5th and 6th ribs, and intercostal muscles) will be observed and a block needle will be directed to the interfacial plane between rhomboid major muscle and intercostal muscle. RIB will be performed by injecting 20 ml of bupivacaine 0.25%. In the same position, the probe will be placed at the midaxillary line at the level of T3, and the landmark points (latissimus dorsi muscle and serratus muscle and intercostal muscles) will be observed. Under sterile conditions, a SAP block will be performed by injecting 20 ml of Bupivacaine 0.25% into the plane between serratus muscle and intercostal muscle.
  Interventions: Procedure: RIB+SAP blocks
- Control Group (No Intervention): No block procedures will be performed in this group.

INTERVENTIONS:
Procedure: RIB+SAP blocks — RIB block will be performed after endotracheal intubation, then a SAP block will be performed. No other intervention will be performed to the patients.
  Arms: Block Group

SUMMARY:
Rhomboid intercostal block is used to block lateral cutaneous branches of intercostal nerves between T3 and T9 dermatomes. Serratus anterior plane block is used to block lateral cutaneous branches of intercostal nerves between T2 and T6, in addition, it is also known to block thoracodorsal nerve and long thoracic nerve. Both of the blocks are usually performed for postoperative analgesia following breast surgery. The primary hypothesis of the study is that FEV1 value of the patients who will receive modified radical mastectomy (MRM) and rhomboid intercostal plane (RIP) block combined with serratus anterior plane (SAP) will be higher than FEV1 value of the patients in the no-block group. The secondary hypothesis is that RIP+SAP blocks will provide reduction in the pain scores and opioid consumption in the postoperative first 24 hours.

DETAILED DESCRIPTION:
The patients who are scheduled for MRM under general anesthesia, aged between 18-65 years and ASA scores I-II will be included in the study. Respiratory functions (FEV₁, FVC, FEV₁/FVC, PEF, FEF25-75) of the patients will be measured by a hand-held spirometry device prior to the operation in the surgical ward. The induction of anesthesia will be provided similarly in all patients, then patients will be intubated and randomly divided into two groups. One group will receive RIP+SAP block using 40 milliliters of %0.25 bupivacaine and patients in the control group will receive no block procedures. The standard analgesia will be provided by intraoperative intravenous (iv) infusion of dexketoprofen 50 mg and iv tramadol 1 mg/kg which will be administered in 15 minutes before end of the surgery. Respiratory functions of the patients will be measured at the postoperative 2nd, 4th and 24th hours. Pain intensity of the patients will be evaluated by Numerical Rating Scale (NRS) which is a scale ranges between 0 (no pain) and 10 (the worst pain that a person can stand). NRS scores will be evaluated at the postoperative 15th, 30th minutes and 1st, 2nd, 6th, 12th and 24th hours, and opioid consumption will be recorded at the postoperative 24th hour.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Female
* Ages between 18-65
* Patients who will receive breast cancer surgery under general anesthesia

Exclusion Criteria:

* Known respiratory diseases
* Rhinitis and atopic dermatitis story
* New York Heart Association Class equal to higher than class 2
* Respiratory diseases story in the last two weeks
* Alchol or substance or chronic opioid consumption story
* Any pain killers intake in the last 24 hours prior to surgery
* Active smokers or ex-smokers
* Body mass index over 35 kg/m2
* İnfection at the injection sites
* Known allergy to local anesthetics
* Known psychiatric diseases
* Operations longer than 3 hours

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | postoperative 2nd hour
  FEV1 of the patients in the block group will be higher at the postoperative second hour than the patients in the control group

SECONDARY OUTCOMES:
Postoperative pain | Postoperative second hour
  The pain scores of the patients in the block group will be lower than the patients in the control group at the postoperative second hour.
Postoperative opioid consumption | Postoperative 24th hour
  The opioid consumption of the patients in the block group will be lower than the patients in the control group at the postoperative 24th hour.
Forced Vital Capacity (FVC) | postoperative 2nd hour
  FVC value of the patients in the block group will be higher at the postoperative second hour than the patients in the control group
FEV1/FVC | postoperative 2nd hour
  FEV1/FVC value of the patients in the block group will be higher at the postoperative second hour than the patients in the control group
forced expiratory flow at 25-75% of forced vital capacity (FEF25-75) | postoperative 2nd hour
  FEF25-75 values of the patients in the block group will be higher at the postoperative second hour than the patients in the control group
Peak expiratory flow (PEF) | postoperative 2nd hour
  PEF values of the patients in the block group will be higher at the postoperative second hour than the patients in the control group

CONTACTS AND LOCATIONS:
Overall Officials: Bakiye Uğur, MD, Study Chair — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with anyone